CLINICAL TRIAL: NCT02174029
Title: Serial Ultrasonographic Evaluation Of Diaphragm Thickness During Mechanical Ventilation In ICU Patients
Brief Title: Serial Daily Diaphragm Ultrasounds in Ventilated Patients
Status: Completed | Type: Observational
Sponsor: Steve Reynolds (Other)
Collaborators: Fraser Health (Other)
Responsible Party: Sponsor-Investigator, Steve Reynolds, Head and Research Director, Department of Critical Care, Royal Columbian Hospital, Fraser Health
Organization: Fraser Health (Other)
Other Study IDs: 2013130
Record Dates: First submitted 2014-05-27; First posted 2014-06-25 (Estimated); Last update posted 2015-03-11 (Estimated); Status verified 2015-03

CONDITIONS: Muscle Atrophy or Weakness; Ventilator-associated Lung Injury
Keywords: Atrophy; Ventilator; Induced; Diaphragm; Dysfunction
MeSH Terms: conditions — Muscular Atrophy; Asthenia; Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Ventilation- mandatory mode only: those patient ventilator days during which they had only received a mandatory mode of ventilation
  Interventions: Procedure: Ventilation- mandatory
- Ventilation- voluntary mode only: Those patient days on a mechanical ventilator who have not received prior mandatory ventilation during this episode of mechanical ventilation.
  Interventions: Procedure: Ventilation- voluntary mode only
- voluntary with preceding mandatory: Those patient ventilator days where the patient had at least one prior day of mandatory mechanical ventilation during this episode of respiratory support.
  Interventions: Procedure: Voluntary with preceding mandatory

INTERVENTIONS:
Procedure: Ventilation- mandatory — Patient days during which only a mandatory ventilation mode was used and prior to this no voluntary mode was used.
  Groups: Ventilation- mandatory mode only
Procedure: Ventilation- voluntary mode only — Patient days on a voluntary mode with no preceding days with a majority of time spend on a mandatory mode
  Groups: Ventilation- voluntary mode only
Procedure: Voluntary with preceding mandatory — Patient days on a voluntary vent mode with at least one day prior during which the majority of the vent mode was mandatory.
  Groups: voluntary with preceding mandatory

SUMMARY:
When a person is put on a breathing machine the investigators think that the breathing muscles can get weaker. The investigators are not sure how quickly this happens but in some people this leads to problems when they try to breathe on their own without the breathing machine. The diaphragm is at the bottom of a person's chest separating their lungs from what is in their belly and it is a very strong muscle. In fact, it is main muscle that one uses for breathing.

An ultrasound machine is a painless way to see what is happening beneath the skin. It is safe and easy to do. Using an ultrasound the investigators are planning to measure how thick the diaphragm is and how much it changes while a person is on a breathing machine in the ICU.

Getting a better understanding of this condition could lead to improved treatments that might help support patients who require a ventilator for breathing.

The investigators hypothesis is that patients for whom the breathing machine is doing all of the work of breathing, will have their diaphragm thickness gradually decrease and changing to a breathing modem mode where they have to put in more effort the diaphragm thickness will start increasing again.

DETAILED DESCRIPTION:
The investigators propose to expand the investigators single-centre longitudinal pilot study into a complete study in which the investigators will use B-mode ultrasonography to evaluate daily changes in diaphragm thickness in all critically ill patients on mechanical ventilation (MV) until successful weaned from MV. The impact of patient age, co-morbidities, and the use of various modes of ventilation on diaphragm thickness will be assessed. Diaphragmatic thickness and its change from baseline will be evaluated as predictors of the need for a prolonged wean (>7days).

The investigators hypothesize that in patients on mandatory mode ventilation, diaphragmatic thickness will progressively decrease. Switching from mandatory to assisted breathing modes will correlate with increases in diaphragmatic thickness.

ELIGIBILITY:
Inclusion Criteria:

* All patients age ≥19 years in the ICU on ventilation

Exclusion Criteria:

* History of diaphragmatic or neuromuscular disease
* On a home ventilator
* History of diaphragm surgery
* Absence of adequate initial US images (3 consecutive days with at least 2 operators)
* BMI greater than 40

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated critical ill patients
Sampling Method: Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2014-06; Primary Completion 2014-08 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
US measurement of diaphragm and quadriceps thickness | Participants will be ultrasounded daily until they are extubated or the 3 month study period has ended, the expected average duration of mechanical ventilation is 4.4 days at our institution
  Diaphragm thickness will be measured once per day and continue until extubation, liberation from mechanical ventilation, transfer to another facility, death, or study completion.

SECONDARY OUTCOMES:
Quadriceps muscle thickness | Participants will be ultrasounded daily until they are extubated or the 3 month study period has ended, the expected average duration of mechanical ventilation is 4.4 days at our institution
  The thickness of the quadriceps muscle on ultrasound will be measured daily until patient exit from study
PEEP (Postive end expiratory pressure) applied by the mechanical ventilator at the time of the ultraspound | Participants will be ultrasounded daily until they are extubated or the 3 month study period has ended, the expected average duration of mechanical ventilation is 4.4 days at our institution
  The PEEP (as described above in the title) in cm H20 as applied by the mechanical ventilator, measured at the time of ultrasound
re-intubated within 48 hours | followed for 48 hours post extubation, or 3 month study period has ended
  Whether a patient required re-intubation within 48 hours of extubation
mean daily fluid balance | Will be recorded daily until they are extubated or the 3 month study period has ended, the expected average duration of mechanical ventilation is 4.4 days at our institution
  Fluid balance of administer fluids minus measurable excreted fluid as recorded every 24 hours by the bedside nurse
mean daily FiO2 (oxygen level administered) | Will be recorded daily until they are extubated or the 3 month study period has ended, the expected average duration of mechanical ventilation is 4.4 days at our institution
  The daily average oxygen delivered through the mechanical ventilator to the patient.
mode of mechanical ventilation for >80% of the day | Will be recorded daily until they are extubated or the 3 month study period has ended, the expected average duration of mechanical ventilation is 4.4 days at our institution
  Mode of mechanical ventilation for the >80% of the day will be recorded here. This will be split into a mandatory mode (where the machine supplies a breath) or a voluntary mode (where the patient triggers the breath and the machine supports it).
steroids given | Will be recorded daily until they are extubated or the 3 month study period has ended, the expected average duration of mechanical ventilation is 4.4 days at our institution
  This will include any dose of steroids administered to the patient each day during their intubation.
vasopressors given | Will be recorded daily until they are extubated or the 3 month study period has ended, the expected average duration of mechanical ventilation is 4.4 days at our institution
  This will include any dose of medications to support the blood pressure (norepinephrine, epinephrine, dopamine, dobutamine, amrinone) administered to the patient each day during their intubation.
paralytics given | Will be recorded daily until they are extubated or the 3 month study period has ended, the expected average duration of mechanical ventilation is 4.4 days at our institution
  This will include any dose of paralytic medication administered to the patient each day during their intubation, except given as part of their initial intubation
30 day mortality | 30 days after patient is extubated, or at the end of the follow up period 1 month after the 3 month study has ended
  This is to capture all cause mortality. A patient will be considered to have survived if they are discharged from hospital.
Body Mass Index (BMI) | from admission information, at the time of admission to the ICU, obtained from the patient record
  The standard BMI will be recorded as determined by the clinical dietician.
presence of sepsis/severe sepsis on admission | from admission information, at the time of admission to the ICU, obtained from the patient record.
  This will be determined as positive if there is any reference to infection in the patients admitting paperwork in conjunction with the classic SIRS (systemic inflammatory response syndrome) criteria.
% Caloric goals met in preceding 24 hours | Will be recorded daily until they are extubated or the 3 month study period has ended, the expected average duration of mechanical ventilation is 4.4 days at our institution
  A % of caloric goals delivered over the preceding 24 hours will be captured
Initial presence of malnutrition | Measure at the time of admission to the ICU
  Presence of malnutrition as assessed by dietician on admission
At risk for re-feeding syndrome | Assessed on admission to the ICU
  Presence of risk for re-feeding syndrome as assessed by dietician on admission

CONTACTS AND LOCATIONS:
Overall Officials: Steven Reynolds, MD, Principal Investigator — Royal Columbian Hospital, Fraser Health
Locations (1):
- Royal Columbian Hospital, New Westminster, British Columbia, Canada